CLINICAL TRIAL: NCT04428632
Title: Expanded Access Program With Oral Berotralstat for the Prevention of Attacks in Patients With Hereditary Angioedema
Brief Title: Oral Berotralstat Expanded Access Program
Status: Approved for marketing | Type: Expanded Access
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: BCX7353-308
Record Dates: First submitted 2020-06-10; First posted 2020-06-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Hereditary Angioedema; HAE; Prophylaxis
Keywords: Berotralstat; BCX7353; Hereditary Angioedema; HAE
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — berotralstat

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Berotralstat — One 150mg capsule administered orally once daily
  Other Names: BCX7353

SUMMARY:
This expanded access program will provide access to berotralstat for eligible participants with hereditary angioedema in the U.S.

DETAILED DESCRIPTION:
Physicians may request access to berotralstat for eligible participants with unmet medical need

Physicians can send email inquiries to access.us@inceptua.com or call 1-888-225-8677

Patients who may be interested should contact their physician about participation

Berotralstat (BCX7353) will be available through this expanded access program until it is commercially available

ELIGIBILITY:
Inclusion Criteria

Patients must meet all of the following inclusion criteria to be eligible for participation in this program:

1. At least 12 years of age
2. Able to provide written, informed consent or assent
3. Patients with a clinical diagnosis of HAE Type I or II who, in the opinion of their treating physician, are expected to benefit from an oral treatment for the prevention of angioedema attacks, and who are not eligible or able to access a berotralstat clinical trial
4. Females must use acceptable effective contraception

Exclusion Criteria

Patients must meet none of the below exclusion criteria to be eligible for participation in this program:

1. Pregnancy or breast-feeding
2. Any clinically significant medical condition or medical history that, in the opinion of the treating physician, would interfere with the patient's safety
3. Current infection with hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult